CLINICAL TRIAL: NCT03567629
Title: A Prospective, Open-lable, Multicenter, Randomized, Controlled Phase II Clinical Trial to Evaluate the Efficacy of Irinotecan Versus Oxaliplatin in the First-line Treatment of Refractory Metastatic Colorectal Cancer
Brief Title: Evaluate the Efficacy of Irinotecan Versus Oxaliplatin in the First-line Treatment of Refractory Metastatic Colorectal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Collaborators: Liaoning Cancer Hospital & Institute (Other); Zhejiang University (Other)
Responsible Party: Principal Investigator, Shen Lin, Head of Head of department of Gastrointestinal oncology, Peking University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSMDT-02
Record Dates: First submitted 2018-06-12; First posted 2018-06-26 (Actual); Last update posted 2018-06-26 (Actual); Status verified 2018-06

CONDITIONS: mCRC
Keywords: Irinotecan; Oxaliplatin; refractory; mCRC
MeSH Terms: interventions — Irinotecan; Fluorouracil; Leucovorin; Capecitabine; S 1 (combination); Bevacizumab; Cetuximab; Oxaliplatin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Irinotecan-based chemotherapy (Experimental)
  Interventions: Drug: Irinotecan
- Oxaliplatin-based chemotherapy (Active Comparator)
  Interventions: Drug: Oxaliplatin

INTERVENTIONS:
Drug: Irinotecan — Irinotecan 180 mg / m2, intravenous drip, D1, combined with fluorouracil / calcium folinate or Capecitabine or S1; combine or not combine with Bevacizumab or Cetuximab; every 14 days for a cycle.
  Other Names: fluorouracil / calcium folinate; Capecitabine; S1; Bevacizumab; Cetuximab
  Arms: Irinotecan-based chemotherapy
Drug: Oxaliplatin — Oxaliplatin 85mg/m2 (two-week regimen) or 130mg/m2 (three week regimen), intravenous drip, D1, combined with fluorouracil / calcium folinate or Capecitabine or S1; combine or not combine with Bevacizumab or Cetuximab; every 14 or 21 days for a cycle.
  Other Names: fluorouracil / calcium folinate; Capecitabine; S1; Bevacizumab; Cetuximab
  Arms: Oxaliplatin-based chemotherapy

SUMMARY:
This is a prospective, open-lable, multicenter, randomized, controlled, phase II clinical study. The aim is to evaluate the efficacy of Irinotecan versus Oxaliplatin in the first-line treatment of refractory metastatic colorectal cancer.

DETAILED DESCRIPTION:
This trial is conducted in patients with the refractory metastatic colorectal cancer. Eligible patients are randomized into two arms at 1:1 ratio to receive Irinotecan-based regimen or Oxaliplatin-based regimen until progress of the disease, unacceptable toxicity or withdrawal of consent by the patient. Study evaluation time is until death of patient or a deadline set by the researchers.

ELIGIBILITY:
Inclusion Criteria:

1. Histopathological diagnosis of metastatic colorectal adenocarcinoma.
2. At least one measurable or assessable lesion that meet RECIST criteria.
3. Accord with standard for refractory colorectal cancer (The standard for refractory colorectal cancer can be met if one of the following conditions is met)

(1) Right colon cancer. (2) Mucinous adenocarcinoma or signet ring cell carcinoma. (3) Complicated by peritoneal metastasis. (4) MSI-H or dMMR, immune checkpoint inhibitor therapy is not acceptable. 4. Male or female, age≥18 years old. 5. Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2. 6. Life expectancy >3 months 7. Adequate organ function as indicated by the following laboratory values:

1. Serum total bilirubin ≤ 1.5 X upper limit of the normal (ULN)
2. Absolute neutrophil count (ANC) ≥1,500 /µL（1.5×109 /L）
3. Platelets ≥100,000 /µL（100×109 /L）
4. Hemoglobin ≥9.0 g/dL
5. Serum creatinine ≤1.5 X (ULN)
6. Prothrombin Time (PT)≤ 1.5 X ULN
7. Left ventricular ejection fraction (LVEF)(measured by Doppler ultrasound) is greater than the lower limit of the normal value (LLN) defined by the study center at which the examination was conducted.

8. Signed the informed consent with name and time. 9. The subjects are accredited with good compliance, and capable to cooperate, completing the relevant examination treatment, and follow-ups.

Exclusion Criteria:

1. Received palliative chemotherapy, such as adjuvant chemotherapy, recurrence within 12 months after adjuvant chemotherapy.
2. Metastatic lesion is subject to be treated by local intervention.
3. Subjects with BRAF V600E mutation.
4. Presence of other active malignancies or a history of other malignancies within the past 5 years, except for carcinoma in situ of the cervix, basal cell carcinoma of the skin that has been previously treated with curative intent.
5. Subjects with cerebral metastasis, spinal cord compression, carcinomatous meningitis, CT /MRI examination reveals diseases of the brain or pia mater during screening.
6. Subjects with chronic diarrhea, intestinal obstruction or incomplete intestinal obstruction, or severe peripheral nerve disease.
7. Any of the following diseases occurred in the 12 months before the study: Myocardial infarction, severe / unstable angina pectoris, coronary artery / peripheral artery bypass grafting, symptomatic congestive heart failure, cerebrovascular accident, or transient ischemic attack, or pulmonary embolism within 6 months
8. Subject is known to be infected with Immunodeficiency virus (HIV) or associated with acquired immune deficiency syndrome (AIDS).
9. Subject is enrolled in other clinical trials currently.
10. Pregnant or lactating women; women of potential childbearing age and male subjects do not use effective contraception during the study period.
11. Other severe acute and chronic physiological or mental problems, or abnormal laboratory tests, which may increase the risk of participating in the study or use of drugs, or interfering with the results of the study, and is judged by the researchers that the patient is not suitable for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Estimated)
Dates: Start 2018-05-29 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival: From date of enrollment until the date of first documented progression or date of death from any cause, whichever came first. | assessed up to 10 months
  Evaluation of the Progression-free Survival of Irinotecan-based regimen versus Oxaliplatin-based regimen in refractory metastatic colorectal cancer patients.

SECONDARY OUTCOMES:
Overall Survival : From date of enrollment until the date of death. | 2 years
  Evaluation of the Overall Survival of Irinotecan-based regimen versus Oxaliplatin-based regimen in refractory metastatic colorectal cancer patients.
Evaluation of PFS in patients with different fluorouracil drugs and different genotyping subgroups. | 10months
  flurouracil drugs：fluorouracil、S1、Capecitabine
Evaluation of OS in patients with different fluorouracil drugs and different genotyping subgroups. | 2 years
  flurouracil drugs：fluorouracil、S1、Capecitabine
The incidence of treatment related emergent adverse events（Safety and Tolerance） | Until 28 days after the deadline of enrollment
  Adverse reactions evaluation is based on the National Cancer Institute adverse event General terminology Standard [CTCAE] 4.0 version

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, Professor, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (1):
- Beijing Cancer Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- Available data/document: Individual Participant Data Set — https://en.wikipedia.org/wiki/United_States_National_Library_of_Medicine